CLINICAL TRIAL: NCT00435227
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate a Single Intramuscular Dose of Motavizumab (MEDI-524), a Humanized Enhanced Potency Monoclonal Antibody Against Respiratory Syncytial Virus (RSV), for the Outpatient Treatment of Children With RSV Illness
Brief Title: A Study to Evaluate a Single Intramuscular Dose of Motavizumab to Treat Children With Respiratory Syncytial Virus (RSV) Illness
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to an inability to enroll the planned number of participants
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MI-CP146
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Participants Less Than 12 Months of Age With RSV Illness
Keywords: Respiratory Syncytial Viruses; RSV
MeSH Terms: interventions — motavizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motavizumab (Experimental): Participants will receive a single IM dose of 30 mg/kg of motavizumab on Day 0 of the study.
  Interventions: Biological: Motavizumab
- Placebo (Placebo Comparator): Participants will receive a single IM dose of placebo matched to motavizumab on Day 0 of the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Motavizumab — A single IM dose of 30 mg/kg will be administered on Day 0 of the study.
  Other Names: MEDI-524
  Arms: Motavizumab
Other: Placebo — A single IM dose of placebo matched to motavizumab will be administered on Day 0 of the study.
  Arms: Placebo

SUMMARY:
This was a Phase 2, randomized, double-blind, placebo-controlled, multicenter study to determine the effect of a single 30 mg/kg intramuscular (IM) dose of motavizumab on viral load and motavizumab levels in the upper respiratory tract of children who present with RSV illness but who do not require hospitalization. Using 1:1 randomization, 30 mg/kg motavizumab or placebo will be administered as soon as possible after a child's diagnosis of RSV and his/her eligibility for the study has been confirmed.

DETAILED DESCRIPTION:
This was a Phase 2, randomized, double-blind, placebo-controlled, multicenter study to determine the effect of a single 30 mg/kg IM dose of motavizumab on viral load in the upper respiratory tract of children who present with RSV illness but who do not require hospitalization. Participants were randomly assigned in a 1:1 ratio to 30 mg/kg motavizumab or placebo as soon as possible after a child's diagnosis of RSV and his/her eligibility for the study had been confirmed. Randomization was stratified by age (<6 months and greater than or equal to 6 to less than or equal to 12 months of age) and by site. Enrollment of an initial 100 children (50 per treatment group) will take place at multiple sites beginning in the 2006-2007 RSV season. The study was terminated early due to inability to enroll the planned number of participants.

ELIGIBILITY:
Inclusion Criteria:

* Previously healthy
* Age ≤12 months at the time of randomization
* Weight ≤10 kg at the time of randomization
* Gestational age ≥36 weeks
* RSV illness (must have coryza) documented by a positive RSV test at the time of evaluation
* Documented stable clinical condition that does not require hospitalization (oxygen saturation ≥ 95%; respiratory rate < 60 breaths/minute in children < 2 months and < 50 breaths/minute in children 2-12 months)
* Respiratory Distress Assessment Instrument (RDAI) score of ≤ 6 (there can be no more than 1 point assigned for each of the 6 assessment categories) at baseline evaluation
* Randomization within 4 hours of being evaluated with a positive Binax® RSV test
* Written informed consent obtained from the participant's parent(s) or legal guardian

Exclusion Criteria:

* Prior receipt of or receiving treatment with steroids (except topical steroids) prior to randomization
* Prior medically diagnosed RSV infection
* Prior receipt of or receiving anti-viral treatment for the current episode of RSV infection prior to randomization
* Any medically significant underlying ongoing chronic illness or organ system dysfunction or other known acute illness, other than the acute RSV infection
* Known renal impairment, hepatic dysfunction, hematologic abnormalities, seizure or other neurologic disorder or immunodeficiency
* Requirement for supplemental oxygen (brief use of oxygen in the immediate postnatal period to treat a transient condition is allowed)
* Mechanical ventilation at any time prior to the onset of the current RSV infection
* Congenital heart disease [children with medically or surgically closed patent ductus arteriosus (PDA), small atrial septal defect (ASD) or small ventricular septal defect (VSD) will be allowed]
* Previous reaction to intravenous immunoglobulin (IVIG), blood products, or other foreign proteins
* Prior use of IVIG, RSV-IGIV (RespiGam®), motavizumab or other immunoglobulin products within the past 2 months
* Prior use of palivizumab (Synagis®) within the past 2 months
* Currently receiving other investigational agents or have received any other investigational agents within the last 3 months
* Prior or current participation in any investigational study with a therapeutic agent or vaccine for RSV

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2007-03-20 (Actual); Primary Completion 2008-05-31 (Actual); Study Completion 2008-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Pamela Griffin, M.D., Study Director — MedImmune LLC
Locations (28):
- United States (28):
  - Research Site, Tucson, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, Paterson, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, The Bronx, New York
  - Research Site, Youngstown, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Richmond, Virginia
  - West Virginia University Pediactric Center, Charleston, West Virginia
  - Research Site, Charleston, West Virginia
  - Research Site, Huntington, West Virginia
  - Research Site, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 20Mar2007 to 31May2008 in the United States of America.
Pre-assignment Details: A total of 12 participants were randomized in the study.
Groups:
- Placebo: Participants received a single intramuscular (IM) dose of placebo matched to motavizumab on Day 0 of the study.
- Motavizumab 30 mg: Participants received a single IM dose of 30 milligrams/kilograms (mg/kg) of motavizumab on Day 0 of the study.
Period: Overall Study
Arm/Group | Placebo | Motavizumab 30 mg
Started | 5 | 7
Completed | 5 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Motavizumab 30 mg | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Continuous [Mean (Standard Deviation); unit: Months] | 3.78 (1.97) | 5.79 (3.68) | 4.95 (3.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Syncytial Virus (RSV) Load in the Upper Respiratory Tract of RSV-infected Participants as Measured by Reverse Transcriptase-polymerase Chain Reaction (RT-PCR) at Day 0
Description: The RSV viral load is measured by real-time RT-PCR in the RSV-infected participants. RSV-infected children are those who are positive for any RSV by RT-PCR of nasal wash aspirates.
Time Frame: Day 0
Population: Intent-to-treat population included all participants who were randomized in the study. Participants who were RSV-positive at Day 0 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 5 | 5
log10 copies/mL | 5.877 (1.503) | 6.657 (0.999)

2. Primary Outcome: RSV Load in the Upper Respiratory Tract of RSV-infected Participants as Measured by RT-PCR at Day 2
Description: as for outcome 1
Time Frame: Day 2
Population: Intent-to-treat population included all participants who were randomized in the study. Participants who were RSV-positive at Day 2 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 5 | 4
log10 copies/mL | 5.070 (1.905) | 5.854 (1.855)

3. Primary Outcome: RSV Load in the Upper Respiratory Tract of RSV-infected Participants as Measured by RT-PCR at Day 30
Description: as for outcome 1
Time Frame: Day 30
Population: Intent-to-treat population included all participants who were randomized in the study. Participants who were RSV-positive at Day 30 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 5 | 5
log10 copies/mL | 2.500 (0.000) | 2.640 (0.312)

4. Primary Outcome: RSV Load in the Upper Respiratory Tract of RSV-infected Participants as Measured by RT-PCR at Day 90
Description: as for outcome 1
Time Frame: Day 90
Population: Intent-to-treat population included all participants who were randomized in the study. Participants who were RSV-positive at Day 90 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 5 | 5
log10 copies/mL | 2.500 (0.000) | 2.500 (0.000)

5. Secondary Outcome: Percentage of Participants Who Have Progression of RSV Illness That Requires Subsequent Hospitalization
Description: The percentage of participants who have progression of RSV illness that requires subsequent hospitalization is reported. RSV illness symptomps included fever, coryza, cough, and parental opinion of return to normal health and activity.
Time Frame: From Randomiation (Day 0) Up to Day 30
Population: Evaluable population for RSV included all participants who were positive for RSV at Study Day 0 as measured by RT-PCR.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 5 | 5
Percentage of participants | 0 | 0

6. Secondary Outcome: Respiratory Assessment Change Score (RACS) Derived From Baseline
Description: The RACS assesses changes in wheezing and retractions as measured by the respiratory distress assessment instrument (RDAI) score and changes in respiratory rate. A RDAI score is a measure of the degree of severity of wheezing and retractions, with score range from 0 to 17; higher scores indicate more severe disease. Respiratory rate is summarized by raw scores and standardized change score. Change in respiratory rate of less than or equal to (<=) 5% from baseline is counted as a change of 0 units and a change in respiratory rate is assigned 1 point per each 10% change in respiratory rate. The RACS is calculated as arithmetic sum of RDAI score change and of the standardized respiratory rate change (for example, a child showing improvement who had a RDAI of -5 and a respiratory rate change of -2 would have a RACS score of -7). The RACS assessment does not have a minimum and/or maximum scale range. A decrease in RACS represents improvement, whereas an increase signifies deterioration.
Time Frame: Baseline (Day 0); and Days 2, 7, and 30
Population: Evaluable population for RSV included all participants who were positive for RSV at Study Day 0 as measured by RT-PCR.
Measure: Mean (Standard Deviation); unit: Units on a score
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 5 | 5
Units on a score
  Day 2 | 1.80 (4.09) | 2.20 (5.81)
  Day 7 | -0.20 (4.82) | -2.00 (1.58)
  Day 30 | -1.40 (4.51) | -2.00 (4.18)

7. Secondary Outcome: Change From Baseline in Oxygen Saturation Level
Description: Change from baseline in oxygen saturation level is reported.
Time Frame: Baseline (Day 0), Days 2, 7, and 30
Population: Evaluable population for RSV included all participants who were positive for RSV at Study Day 0 as measured by RT-PCR.
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 5 | 5
Percentage of oxygen saturation
  Day 2 | 1.00 (1.73) | -1.00 (1.58)
  Day 7 | 1.20 (2.17) | 0.60 (1.34)
  Day 30 | 1.80 (1.48) | 0.40 (1.52)

8. Secondary Outcome: Change in RACS of RSV-infected Outpatient Participants Who Subsequently Required Hospitalization
Description: The RACS assesses changes in wheezing and retractions as measured by the RDAI score and changes in respiratory rate. A RDAI score is a measure of the degree of severity of wheezing and retractions, with score range from 0 to 17; higher scores indicate more severe disease. Respiratory rate is summarized by raw scores and standardized change score. A change in respiratory rate of <= 5% from baseline is counted as a change of 0 units and a change in respiratory rate is assigned 1 point per each 10% change in the respiratory rate. The RACS is calculated as the arithmetic sum of the RDAI score change and of the standardized respiratory rate change (for example, a child showing improvement who had a RDAI of -5 and a respiratory rate change of -2 would have a RACS score of -7). The RACS assessment does not have a minimum and/or maximum scale range. A decrease in the RACS represents improvement, whereas an increase signifies deterioration.
Time Frame: Baseline (Day 0) to Day 30
Population: Evaluable population for RSV included all participants who were positive for RSV at Study Day 0 as measured by RT-PCR. Data were not collected as no participants required hospitalization.
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Oxygen Saturation Levels in RSV-infected Outpatient Participants Who Subsequently Required Hospitalization
Time Frame: Baseline (Day 0) to Day 30
Population: as for outcome 8
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Heart Rate of RSV-infected Outpatient Participants Who Subsequently Required Hospitalization
Time Frame: Baseline (Day 0) to Day 30
Population: as for outcome 8
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Respiratory Rate of RSV-infected Outpatient Participants Who Subsequently Required Hospitalization
Time Frame: Baseline (Day 0) to Day 30
Population: as for outcome 8
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants Who Required Hospitalization, Intensive Care Unit (ICU) Stay, Supplemental Oxygen, and Mechanical Ventilation
Description: Number of participants who required hospitalization, ICU stay, supplemental oxygen, and mechanical ventilation is reported.
Time Frame: Baseline (Day 0) to Day 90
Population: Evaluable population for RSV included all participants who were positive for RSV at Study Day 0 as measured by RT-PCR.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 5 | 5
Participants
  Hospitalization | 0 | 0
  Supplemental oxygen | 0 | 0
  Mechanical ventilation | 0 | 0
  ICU stay | 0 | 0

13. Secondary Outcome: Duration of Hospitalization, ICU Stay, Supplemental Oxygen Used, and Mechanical Ventilation Required
Time Frame: Baseline (Day 0) to Day 90
Population: Evaluable population for RSV included all participants who were positive for RSV at Study Day 0 as measured by RT-PCR. Data were not collected as no participants were hospitalized or received intensive care or supplemental oxygen, or mechanical ventilation.
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Number of Participants Who Progresses From Upper Respiratory Tract Infection to Lower Respiratory Tract Infection (LRI)
Description: A LRI event is one that has a medical diagnosis of bronchiolitis or pneumonia. In the absence of such a medical diagnosis, the occurrence of LRI events will be determined by the principal investigator after review of the medical record and based on the presence of retractions or lower respiratory tract rhonchi, wheezing, crackles, or rales in children with a positive RSV test.
Time Frame: Baseline (Day 0) to Day 30
Population: Safety population included all participants who had received any study drug and had any follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 5 | 7
Participants | 0 | 1

15. Secondary Outcome: Number of LRI Infected Participants Who Required Hospitalization, ICU Stay, Supplemental Oxygen, Mechanical Ventilation, and Respiratory Medications
Description: Number of LRI infected participants who required hospitalization, ICU stay, supplemental oxygen, mechanical ventilation, and respiratory medications are reported.
Time Frame: Baseline (Day 0) to Day 30
Population: Safety population included all participants who had received any study drug and had any follow-up. Participants with LRI were analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 0 | 1
Participants
  Hospitalization | 0 | 0
  Supplemental oxygen | 0 | 0
  Mechanical ventilation | 0 | 0
  ICU stay | 0 | 0
  Respiratory medication | 0 | 0

16. Secondary Outcome: RACS in Participants With LRI
Description: The RACS assesses changes in wheezing and retractions as measured by RDAI score and changes in respiratory rate. A RDAI score is a measure of degree of severity of wheezing and retractions, with score range from 0 to 17; higher scores indicate more severe disease. Respiratory rate is summarized by raw scores and standardized change score. A change in respiratory rate of <= 5% from baseline is counted as a change of 0 units and a change in respiratory rate is assigned 1 point per each 10% change in the respiratory rate. The RACS is calculated as the arithmetic sum of the RDAI score change and of the standardized respiratory rate change (for example, a child showing improvement who had a RDAI of -5 and a respiratory rate change of -2 would have a RACS score of -7). The RACS assessment does not have a minimum and/or maximum scale range. A decrease in the RACS represents improvement, whereas an increase signifies deterioration. RACS in participants with LRI is reported.
Time Frame: From Baseline (Day 0) to Days 2, 7, and 30
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Units on a score
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 0 | 1
Units on a score
  Day 2 |  | 12 (NA) — Standard deviation data was not applicable as only one participant was evaluable for the specified outcome measure.
  Day 7 |  | -4 (NA) — Standard deviation data was not applicable as only one participant was evaluable for the specified outcome measure.
  Day 30 |  | -1 (NA) — Standard deviation data was not applicable as only one participant was evaluable for the specified outcome measure.

17. Secondary Outcome: Motavizumab Concentration in Upper Respiratory Tract
Description: Motavizumab concentration in upper respiratory tract (nasal wash aspirates) is reported.
Time Frame: Days 0 (pre-dose), 2, and 30
Population: Evaluable population for pharmacokinetic (PK) included all participants who have received a full dose of study drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Motavizumab 30 mg
Number analyzed (Participants) | 7
ng/mL
  Day 0 | NA (NA) — The data was not reported as the concentration was below the level of detection.
  Day 2 | 1216.186 (1828.934)
  Day 30 | 348.256 (507.979)

18. Secondary Outcome: Serum Concentration of Motavizumab
Description: Serum concentration of motavizumab is reported.
Time Frame: Days 2, 30, and 90
Population: Evaluable population for PK included all participants who have received a full dose of study drug.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Motavizumab 30 mg
Number analyzed (Participants) | 7
mcg/mL
  Day 2 | 216.761 (43.867)
  Day 30 | 126.296 (25.013)
  Day 90 | 23.799 (9.810)

19. Secondary Outcome: Numbers of Participants With Positive Anti-Motavizumab Antibodies
Description: The number of participants with positive serum antibodies to motavizumab are reported.
Time Frame: Days 0 (pre-dose) and 90
Population: Evaluable population for ADA included all participants who have received a full dose of study drug. Participants with adequate ADA samples were analysed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Motavizumab 30 mg
Number analyzed (Participants) | 7
Participants
  Day 0: number analyzed (Participants) | 6
  Day 0 | 0
  Day 90 | 0

20. Secondary Outcome: Serum Cytokine Levels
Description: Serum Cytokine Levels are reported.
Time Frame: Days 0 (pre-dose), 30, and 90
Population: Evaluable population for RSV included all participants who were positive for RSV at Study Day 0 as measured by RT-PCR. Participants with adequate cytokine levels at specified time points were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: Picograms per millilitre (pg/mL)
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 5 | 5
Picograms per millilitre (pg/mL)
  Interleukin 1 (IL-1) beta: Day 0: number analyzed (Participants) | 5 | 4
  Interleukin 1 (IL-1) beta: Day 0 | 8.000 (0.000) | 8.000 (0.000)
  IL-1 beta: Day 30: number analyzed (Participants) | 4 | 5
  IL-1 beta: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  IL-1 beta: Day 90: number analyzed (Participants) | 4 | 5
  IL-1 beta: Day 90 | 8.000 (0.000) | 8.000 (0.000)
  IL-1 receptor antagonist (RA): Day 0: number analyzed (Participants) | 5 | 4
  IL-1 receptor antagonist (RA): Day 0 | 8.000 (0.000) | 8.000 (0.000)
  IL-1 RA: Day 30: number analyzed (Participants) | 4 | 5
  IL-1 RA: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  IL-1 RA: Day 90: number analyzed (Participants) | 4 | 5
  IL-1 RA: Day 90 | 11.000 (6.000) | 10.960 (6.619)
  IL-2: Day 0: number analyzed (Participants) | 5 | 4
  IL-2: Day 0 | 8.000 (0.000) | 8.000 (0.000)
  IL-2: Day 30: number analyzed (Participants) | 4 | 5
  IL-2: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  IL-2: Day 90: number analyzed (Participants) | 4 | 5
  IL-2: Day 90 | 8.000 (0.000) | 8.000 (0.000)
  IL-4: Day 0: number analyzed (Participants) | 5 | 4
  IL-4: Day 0 | 8.000 (0.000) | 8.000 (0.000)
  IL-4: Day 30: number analyzed (Participants) | 4 | 5
  IL-4: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  IL-4: Day 90: number analyzed (Participants) | 4 | 5
  IL-4: Day 90 | 10.900 (5.800) | 13.060 (11.315)
  IL-5: Day 0: number analyzed (Participants) | 5 | 4
  IL-5: Day 0 | 1.600 (0.000) | 1.600 (0.000)
  IL-5: Day 30: number analyzed (Participants) | 4 | 5
  IL-5: Day 30 | 1.600 (0.000) | 1.600 (0.000)
  IL-5: Day 90: number analyzed (Participants) | 4 | 5
  IL-5: Day 90 | 19.925 (35.460) | 3.080 (3.309)
  IL-6: Day 0: number analyzed (Participants) | 5 | 4
  IL-6: Day 0 | 2.620 (2.281) | 12.025 (8.247)
  IL-6: Day 30: number analyzed (Participants) | 4 | 5
  IL-6: Day 30 | 1.600 (0.000) | 1.980 (0.850)
  IL-6: Day 90: number analyzed (Participants) | 4 | 5
  IL-6: Day 90 | 22.950 (16.093) | 4.040 (3.335)
  IL-7: Day 0: number analyzed (Participants) | 5 | 4
  IL-7: Day 0 | 8.000 (0.000) | 8.000 (0.000)
  IL-7: Day 30: number analyzed (Participants) | 4 | 5
  IL-7: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  IL-7: Day 90: number analyzed (Participants) | 4 | 5
  IL-7: Day 90 | 8.000 (0.000) | 8.000 (0.000)
  IL-8: Day 0: number analyzed (Participants) | 5 | 4
  IL-8: Day 0 | 28.500 (1.728) | 28.525 (14.061)
  IL-8: Day 30: number analyzed (Participants) | 4 | 5
  IL-8: Day 30 | 12.900 (4.678) | 7.900 (2.904)
  IL-8: Day 90: number analyzed (Participants) | 4 | 5
  IL-8: Day 90 | 38.475 (43.752) | 12.120 (4.727)
  IL-9: Day 0: number analyzed (Participants) | 5 | 4
  IL-9: Day 0 | 1.600 (0.000) | 1.600 (0.000)
  IL-9: Day 30: number analyzed (Participants) | 4 | 5
  IL-9: Day 30 | 1.600 (0.000) | 3.020 (3.175)
  IL-9: Day 90: number analyzed (Participants) | 4 | 5
  IL-9: Day 90 | 7.925 (6.758) | 4.200 (4.591)
  IL-10: Day 0: number analyzed (Participants) | 5 | 4
  IL-10: Day 0 | 36.400 (28.205) | 29.625 (31.852)
  IL-10: Day 30: number analyzed (Participants) | 4 | 5
  IL-10: Day 30 | 19.325 (13.297) | 8.000 (0.000)
  IL-10: Day 90: number analyzed (Participants) | 4 | 5
  IL-10: Day 90 | 13.900 (7.161) | 8.000 (0.000)
  IL-11: Day 0: number analyzed (Participants) | 3 | 1
  IL-11: Day 0 | 13.133 (5.860) | 9.750 (NA) — Standard deviation is not applicable as only one participant was evaluable for the specified time point.
  IL-11: Day 30: number analyzed (Participants) | 3 | 3
  IL-11: Day 30 | 15.600 (10.132) | 27.000 (29.878)
  IL-11: Day 90: number analyzed (Participants) | 3 | 3
  IL-11: Day 90 | 148.483 (143.545) | 38.783 (32.632)
  IL-12 P70: Day 0: number analyzed (Participants) | 5 | 4
  IL-12 P70: Day 0 | 8.000 (0.000) | 8.000 (0.000)
  IL-12 P70: Day 30: number analyzed (Participants) | 4 | 5
  IL-12 P70: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  IL-12 P70: Day 90: number analyzed (Participants) | 4 | 5
  IL-12 P70: Day 90 | 20.450 (24.900) | 8.000 (0.000)
  IL-13: Day 0: number analyzed (Participants) | 5 | 4
  IL-13: Day 0 | 8.000 (0.000) | 8.000 (0.000)
  IL-13: Day 30: number analyzed (Participants) | 4 | 5
  IL-13: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  IL-13: Day 90: number analyzed (Participants) | 4 | 5
  IL-13: Day 90 | 8.000 (0.000) | 11.060 (6.842)
  IL-15: Day 0: number analyzed (Participants) | 5 | 4
  IL-15: Day 0 | 1.600 (0.000) | 1.600 (0.000)
  IL-15: Day 30: number analyzed (Participants) | 4 | 5
  IL-15: Day 30 | 1.600 (0.000) | 1.600 (0.000)
  IL-15: Day 90: number analyzed (Participants) | 4 | 5
  IL-15: Day 90 | 2.100 (1.000) | 1.600 (0.000)
  IL-17: Day 0: number analyzed (Participants) | 5 | 4
  IL-17: Day 0 | 2.160 (1.252) | 1.600 (0.000)
  IL-17: Day 30: number analyzed (Participants) | 4 | 5
  IL-17: Day 30 | 2.675 (2.150) | 1.600 (0.000)
  IL-17: Day 90: number analyzed (Participants) | 4 | 5
  IL-17: Day 90 | 29.875 (37.289) | 5.180 (6.324)
  Eotaxin: Day 0: number analyzed (Participants) | 5 | 4
  Eotaxin: Day 0 | 120.860 (53.095) | 116.325 (15.866)
  Eotaxin: Day 30: number analyzed (Participants) | 4 | 5
  Eotaxin: Day 30 | 117.500 (54.553) | 105.720 (19.212)
  Eotaxin: Day 90: number analyzed (Participants) | 4 | 5
  Eotaxin: Day 90 | 139.275 (32.062) | 87.960 (29.430)
  Interferon (IFN) gamma: Day 0: number analyzed (Participants) | 5 | 4
  Interferon (IFN) gamma: Day 0 | 16.020 (10.991) | 8.000 (0.000)
  IFN gamma: Day 30: number analyzed (Participants) | 4 | 5
  IFN gamma: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  IFN gamma: Day 90: number analyzed (Participants) | 4 | 5
  IFN gamma: Day 90 | 115.675 (125.181) | 14.740 (10.698)
  IFN alpha 2: Day 0: number analyzed (Participants) | 5 | 4
  IFN alpha 2: Day 0 | 8.000 (0.000) | 12.000 (8.000)
  IFN alpha 2: Day 30: number analyzed (Participants) | 4 | 5
  IFN alpha 2: Day 30 | 8.000 (0.000) | 12.060 (9.078)
  IFN alpha 2: Day 90: number analyzed (Participants) | 4 | 5
  IFN alpha 2: Day 90 | 20.175 (24.350) | 12.220 (5.792)
  IFN gamma induced protein (IP)-10: Day 0: number analyzed (Participants) | 5 | 4
  IFN gamma induced protein (IP)-10: Day 0 | 605.740 (299.105) | 723.950 (442.489)
  IP-10: Day 30: number analyzed (Participants) | 4 | 5
  IP-10: Day 30 | 518.775 (617.131) | 136.360 (59.356)
  IP-10: Day 90: number analyzed (Participants) | 4 | 5
  IP-10: Day 90 | 310.150 (154.371) | 287.000 (58.101)
  Monocyte Chemoattractant Protein-1 (MCP-1): Day 0: number analyzed (Participants) | 5 | 4
  Monocyte Chemoattractant Protein-1 (MCP-1): Day 0 | 729.860 (248.023) | 717.850 (585.336)
  MCP-1: Day 30: number analyzed (Participants) | 4 | 5
  MCP-1: Day 30 | 728.225 (245.660) | 727.620 (635.702)
  MCP-1: Day 90: number analyzed (Participants) | 4 | 5
  MCP-1: Day 90 | 596.125 (154.409) | 542.320 (294.697)
  Macrophage inflammatory protein (MIP)-1 alpha:Day0: number analyzed (Participants) | 5 | 4
  Macrophage inflammatory protein (MIP)-1 alpha:Day0 | 8.000 (0.000) | 8.000 (0.000)
  MIP-1 alpha:Day 30: number analyzed (Participants) | 4 | 5
  MIP-1 alpha:Day 30 | 10.000 (4.000) | 8.000 (0.000)
  MIP-1 alpha: Day 90: number analyzed (Participants) | 4 | 5
  MIP-1 alpha: Day 90 | 25.375 (15.504) | 8.000 (0.000)
  MIP-1 beta: Day 0: number analyzed (Participants) | 5 | 4
  MIP-1 beta: Day 0 | 99.560 (40.959) | 70.150 (40.912)
  MIP-1 beta: Day 30: number analyzed (Participants) | 4 | 5
  MIP-1 beta: Day 30 | 92.513 (52.444) | 95.700 (58.140)
  MIP-1 beta: Day 90: number analyzed (Participants) | 4 | 5
  MIP-1 beta: Day 90 | 117.300 (43.226) | 77.780 (39.844)
  Rantes: Day 0: number analyzed (Participants) | 5 | 3
  Rantes: Day 0 | 23103.400 (10200.333) | 35348.767 (11488.336)
  Rantes: Day 30: number analyzed (Participants) | 4 | 5
  Rantes: Day 30 | 26038.788 (3942.021) | 29950.000 (13143.128)
  Rantes: Day 90: number analyzed (Participants) | 4 | 5
  Rantes: Day 90 | 41813.725 (45065.022) | 30770.200 (15335.152)
  TNF alpha: Day 0: number analyzed (Participants) | 5 | 4
  TNF alpha: Day 0 | 25.320 (9.373) | 23.075 (4.802)
  TNF alpha: Day 30: number analyzed (Participants) | 4 | 5
  TNF alpha: Day 30 | 21.925 (7.509) | 21.200 (5.482)
  TNF alpha: Day 90: number analyzed (Participants) | 4 | 5
  TNF alpha: Day 90 | 21.925 (6.879) | 21.040 (6.474)
  Soluble IL-2 receptor (SIL-2R) alpha: Day 0: number analyzed (Participants) | 5 | 4
  Soluble IL-2 receptor (SIL-2R) alpha: Day 0 | 116.500 (81.702) | 165.425 (78.977)
  sIL-2R alpha: Day 30: number analyzed (Participants) | 4 | 5
  sIL-2R alpha: Day 30 | 117.988 (93.112) | 108.060 (49.831)
  SIL-2R alpha: Day 90: number analyzed (Participants) | 4 | 5
  SIL-2R alpha: Day 90 | 72.325 (12.848) | 84.060 (48.465)

21. Secondary Outcome: Nasal Wash Cytokine Levels
Description: Nasal wash cytokine levels are reported.
Time Frame: Days 0 (pre-dose), 2, 30, and 90
Population: Evaluable population for RSV included all participants who were positive for RSV at Study Day 0 as measured by RT-PCR. Participants with adequate nasal wash cytokine levels at specified time points were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 5 | 5
pg/mL
  IL-1 beta: Day 0 | 79.380 (164.902) | 282.380 (355.694)
  IL-1 beta: Day 2: number analyzed (Participants) | 4 | 3
  IL-1 beta: Day 2 | 94.050 (123.565) | 144.367 (113.883)
  IL-1 beta: Day 30 | 10.520 (19.946) | 156.240 (336.673)
  IL-1 beta: Day 90 | 4.300 (4.391) | 2.680 (2.415)
  IL-1 RA: Day 0 | 79.200 (88.851) | 205.040 (249.143)
  IL-1 RA: Day 2: number analyzed (Participants) | 4 | 3
  IL-1 RA: Day 2 | 69.225 (50.434) | 255.533 (184.664)
  IL-1 RA: Day 30 | 38.460 (68.111) | 94.600 (123.754)
  IL-1 RA: Day 90 | 24.100 (22.976) | 39.240 (30.922)
  IL-2: Day 0 | 8.000 (0.000) | 8.000 (0.000)
  IL-2: Day 2: number analyzed (Participants) | 4 | 3
  IL-2: Day 2 | 8.000 (0.000) | 8.000 (0.000)
  IL-2: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  IL-4: Day 0 | 25.820 (34.379) | 14.160 (13.774)
  IL-4: Day 2: number analyzed (Participants) | 4 | 3
  IL-4: Day 2 | 8.000 (0.000) | 22.300 (17.419)
  IL-4: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  IL-4: Day 90 | 36.120 (29.029) | 8.000 (0.000)
  IL-5: Day 0 | 1.600 (0.000) | 1.600 (0.000)
  IL-5: Day 2: number analyzed (Participants) | 4 | 3
  IL-5: Day 2 | 1.600 (0.000) | 1.600 (0.000)
  IL-5: Day30 | 1.600 (0.000) | 1.600 (0.000)
  IL-5: Day 90 | 1.600 (0.000) | 1.600 (0.000)
  IL-6: Day 0 | 172.480 (327.548) | 411.320 (477.909)
  IL-6: Day 2: number analyzed (Participants) | 4 | 3
  IL-6: Day 2 | 42.950 (28.197) | 278.467 (231.477)
  IL-6: Day 30 | 3.300 (3.801) | 19.440 (21.978)
  IL-6: Day 90 | 6.540 (7.079) | 7.300 (6.300)
  IL-7: Day 0 | 15.220 (7.083) | 19.480 (12.696)
  IL-7: Day 2: number analyzed (Participants) | 4 | 3
  IL-7: Day 2 | 15.700 (8.895) | 30.567 (10.058)
  IL-7: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  IL-7: Day 90 | 13.460 (7.537) | 11.620 (8.095)
  IL-8: Day 0 | 701.600 (746.108) | 1488.540 (791.215)
  IL-8: Day 2: number analyzed (Participants) | 4 | 3
  IL-8: Day 2 | 1347.975 (760.276) | 2000.000 (0.000)
  IL-8: Day 30 | 424.040 (881.148) | 942.360 (976.506)
  IL-8: Day 90 | 126.260 (151.768) | 312.760 (269.980)
  IL-9: Day 0 | 1.600 (0.000) | 1.920 (0.716)
  IL-9: Day 2: number analyzed (Participants) | 4 | 3
  IL-9: Day 2 | 2.525 (1.850) | 4.400 (3.208)
  IL-9: Day 30 | 1.600 (0.000) | 1.600 (0.000)
  IL-9: Day 90 | 1.600 (0.000) | 1.600 (0.000)
  IL-10: Day 0 | 54.660 (94.235) | 36.840 (31.400)
  IL-10: Day 2: number analyzed (Participants) | 4 | 3
  IL-10: Day 2 | 34.650 (55.865) | 115.867 (123.508)
  IL-10 Day 30 | 3.180 (3.533) | 15.340 (20.013)
  IL-10: Day 90 | 4.700 (4.699) | 2.820 (2.728)
  IL-11: Day 0: number analyzed (Participants) | 5 | 4
  IL-11: Day 0 | 9.750 (0.000) | 9.750 (0.000)
  IL-11: Day 2: number analyzed (Participants) | 4 | 2
  IL-11: Day 2 | 9.750 (0.000) | 9.750 (0.000)
  IL-11: Day 30: number analyzed (Participants) | 5 | 4
  IL-11: Day 30 | 9.750 (0.000) | 9.750 (0.000)
  IL-11: Day 90: number analyzed (Participants) | 5 | 4
  IL-11: Day 90 | 9.750 (0.000) | 9.750 (0.000)
  IL-12 P70: Day 0 | 11.380 (7.558) | 10.240 (5.009)
  IL-12 P70: Day 2: number analyzed (Participants) | 4 | 3
  IL-12 P70: Day 2 | 8.000 (0.000) | 10.967 (5.138)
  IL-12 P70: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  IL-12 P70: Day 90 | 8.000 (0.000) | 8.000 (0.000)
  IL-13: Day 0 | 8.000 (0.000) | 8.000 (0.000)
  IL-13: Day 2: number analyzed (Participants) | 4 | 3
  IL-13: Day 2 | 8.000 (0.000) | 11.033 (5.254)
  IL-13: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  IL-13: Day 90 | 8.000 (0.000) | 8.000 (0.000)
  IL-15: Day 0 | 2.900 (2.907) | 6.580 (4.089)
  IL-15: Day 2: number analyzed (Participants) | 4 | 3
  IL-15: Day 2 | 3.275 (2.311) | 7.900 (1.418)
  IL-15: Day 30 | 1.600 (0.000) | 2.580 (1.470)
  IL-15: Day 90 | 1.960 (0.805) | 2.300 (1.565)
  IL-17: Day 0 | 2.640 (2.326) | 3.060 (2.024)
  IL-17: Day 2: number analyzed (Participants) | 4 | 3
  IL-17: Day 2 | 2.475 (1.750) | 2.900 (2.252)
  IL-17: Day 30 | 1.600 (0.000) | 1.600 (0.000)
  IL-17: Day 90 | 1.980 (0.850) | 1.600 (0.000)
  Eotaxin: Day 0 | 14.500 (10.201) | 20.620 (8.461)
  Eotaxin: Day 2: number analyzed (Participants) | 4 | 3
  Eotaxin: Day 2 | 17.625 (11.507) | 29.300 (7.758)
  Eotaxin: Day 30 | 10.280 (5.098) | 15.420 (11.445)
  Eotaxin: Day 90 | 10.940 (6.574) | 10.540 (5.680)
  IFN gamma: Day 0 | 6.740 (11.493) | 5.760 (2.788)
  IFN gamma: Day 2: number analyzed (Participants) | 4 | 3
  IFN gamma: Day 2 | 4.750 (5.170) | 9.433 (4.140)
  IFN gamma: Day 30 | 1.600 (0.000) | 1.600 (0.000)
  IFN gamma: Day 90 | 1.940 (0.760) | 2.080 (1.073)
  IFN alpha 2: Day 0 | 11.580 (8.005) | 16.900 (8.306)
  IFN alpha 2: Day 2: number analyzed (Participants) | 4 | 3
  IFN alpha 2: Day 2 | 12.075 (8.150) | 19.800 (11.377)
  IFN alpha 2: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  IFN alpha 2: Day 90 | 11.480 (4.774) | 11.220 (7.200)
  IP-10: Day 0 | 3030.820 (3653.453) | 5850.060 (4510.860)
  IP-10: Day 2: number analyzed (Participants) | 4 | 3
  IP-10: Day 2 | 2699.550 (3369.371) | 4405.733 (4604.409)
  IP-10: Day 30: number analyzed (Participants) | 4 | 5
  IP-10: Day 30 | 40.000 (0.000) | 1378.140 (1435.513)
  IP-10: Day 90 | 148.980 (90.285) | 344.720 (201.758)
  MCP-1: Day 0 | 138.280 (261.810) | 352.860 (400.479)
  MCP-1: Day 2: number analyzed (Participants) | 4 | 3
  MCP-1: Day 2 | 67.950 (72.134) | 204.000 (239.883)
  MCP-1: Day 30 | 15.160 (16.010) | 75.900 (69.833)
  MCP-1: Day 90 | 13.580 (7.651) | 30.580 (21.161)
  MIP-1 alpha: Day 0 | 229.060 (463.273) | 116.280 (109.432)
  MIP-1 alpha: Day 2: number analyzed (Participants) | 4 | 3
  MIP-1 alpha: Day 2 | 96.875 (102.773) | 63.300 (57.022)
  MIP-1 alpha: Day 30 | 34.720 (59.748) | 83.880 (118.987)
  MIP-1 alpha: Day 90 | 15.420 (16.592) | 8.000 (0.000)
  MIP-1 beta: Day 0 | 113.840 (211.563) | 88.340 (91.090)
  MIP-1 beta: Day 2: number analyzed (Participants) | 4 | 3
  MIP-1 beta: Day 2 | 74.850 (53.517) | 54.467 (30.928)
  MIP-1 beta: Day 30 | 18.480 (23.434) | 47.700 (71.854)
  MIP-1 beta: Day 90 | 14.560 (14.669) | 10.480 (5.545)
  Rantes: Day 0 | 197.860 (404.890) | 56.720 (72.686)
  Rantes: Day 2: number analyzed (Participants) | 4 | 3
  Rantes: Day 2 | 23.400 (15.609) | 90.067 (116.383)
  Rantes: Day 30: number analyzed (Participants) | 4 | 5
  Rantes: Day 30 | 1.600 (0.000) | 60.560 (97.653)
  Rantes: Day 90 | 4.260 (3.717) | 5.140 (5.594)
  TNF alpha: Day 0 | 104.180 (222.984) | 133.220 (122.334)
  TNF alpha: Day 2: number analyzed (Participants) | 4 | 3
  TNF alpha: Day 2 | 29.425 (30.522) | 44.133 (34.563)
  TNF alpha: Day 30 | 3.440 (4.114) | 22.340 (32.064)
  TNF alpha: Day 90 | 3.980 (5.322) | 2.020 (0.939)
  SIL-2R alpha: Day 0 | 10.500 (5.590) | 14.580 (9.265)
  SIL-2R alpha: Day 2: number analyzed (Participants) | 4 | 3
  SIL-2R alpha: Day 2 | 10.000 (4.000) | 13.167 (8.949)
  SIL-2R alpha: Day 30: number analyzed (Participants) | 4 | 5
  SIL-2R alpha: Day 30 | 8.000 (0.000) | 8.000 (0.000)
  SIL-2R alpha: Day 90 | 8.000 (0.000) | 8.000 (0.000)
  IL-2: Day 90 | 8.000 (0.000) | 8.000 (0.000)

22. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: From the administration of study drug (Day 0) through Day 90
Population: Safety population included all participants who had received any study drug and had any follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab 30 mg
Number analyzed (Participants) | 5 | 7
Participants
  TEAEs | 5 | 6
  TESAEs | 2 | 0

ADVERSE EVENTS:
Time Frame: From the administration of study drug (Day 0) through Day 90
Arm/Group | Placebo | Motavizumab 30 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/7
Other Adverse Events (participants affected / at risk) | 5/5 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5) | Motavizumab 30 mg (N=7)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=5) | Motavizumab 30 mg (N=7)
Conjunctivitis (Eye disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 1 (1)
Teething (Gastrointestinal disorders) | 1 (1) | 3 (3)
Irritability (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 3 (4) | 3 (3)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Viral skin infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Feeding disorder of infancy or early childhood (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2)
Heat rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
On 21Feb2008, the study was terminated earlier than planned completion time due to an inability to enroll planned number of participants. Due to low enrollment, the data for outcome measure of "Duration of symptoms of RSV illness" was not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.